CLINICAL TRIAL: NCT01666249
Title: Evaluation of the Clinic Efficacy of Immunoglobulin Anti-RhD KamRho-D® (Panamerican) in Postpartum Immunization of Rh and Coombs Negative Women at Sensitization Risk.
Brief Title: Clinical Efficacy of Postpartum Immunization of Rh and Coombs Negative Women With Sensitization Risk.
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Suspended for indetermined period.
Sponsor: Azidus Brasil (Industry)
Collaborators: Panamerican Medical Supply (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IMUPAN1011; Emenda 3.0 - 19/09/2017 (Other: Azidus Brasil Pesquisa Científica e Desenvolvimento Ltda.)
Record Dates: First submitted 2012-07-25; First posted 2012-08-16 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy; Fetomaternal Hemorrhage
Keywords: FMH; anti-Rh; efficacy
MeSH Terms: conditions — Fetomaternal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunoglobulin Anti-RhD (Experimental): Participants will receive a single intramuscular administration of 300 mcg/2mL, correponding 1500 UI of Human Immunoglobulin Anti-RhD (Kamrho-D - Panamerican), up to 72 hours post exposition (child-birth).
  Interventions: Biological: Immunoglobulin Anti-RhD

INTERVENTIONS:
Biological: Immunoglobulin Anti-RhD — Participants will receive a single intramuscular administration of 300 mcg/2mL, correponding 1500 UI of Human Immunoglobulin Anti-RhD (Kamrho-D - Panamerican), up to 72 hours post exposition (child-birth).
  Other Names: KamRho-D

SUMMARY:
This a open, prospective, multicenter, single-arm, phase III study for clinical assessment of anti-Rh immunoglobulin (KamRho-D®) in Rh and Coombs negative women with risk sensitization. The anti-Rh immunoglobulin is an immunobiological containing high concentration of specific antibodies against factor D and "neutralizes" D antigen present in the Rh-positive fetal red blood cells (Rh +), which passed into the bloodstream of Rh-negative pregnant women (Rh).

DETAILED DESCRIPTION:
This a phase III study in which women participants with RH and Coombs negative will receive only one dose of 1500 IU anti-Rh immunoglobulin intramuscularly up to 72 hours post exposition (child-birth) and will be following until six months to verification of negative Coombs maintenance. Safety evaluation data will include report of all adverse events (including type, frequency, intensity, seriousness, severity and action taken related to the investigational product).

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate, sign and date ICF;
* 18 years old or older;
* Mothers who are Rh-negative, negative indirect Coombs analyzed by gel agglutination method, whose just deliveries Rh positive baby.

Exclusion Criteria:

* Be participating simultaneously or have participated in another clinical trial within the last 12 months;
* Mothers who are allergic to any components of the formula;
* Mothers who have a history of IgA deficiency or IgA antibody present;
* Mothers who have a history of autoimmune hemolytic anemia with hemolysis or with pre-existing risk of hemolysis;
* Mothers who have indirect Coombs test positive at the beginning of the treatment;
* Rh-negative mothers whose delivered Rh-negative babies;
* Abnormalities of the coagulation system;
* Patients who made use of vaccines made with live pathogens in the last 03 months or will make during the study;
* Patients with clinical diagnosis of prenatal liver and / or severe nephropathy;
* Principal Investigator of the study criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 347 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2020-12

PRIMARY OUTCOMES:
Negative result for coombs test up to six months after immunization | up to six months
  Will be evaluated by proportion of participants that presented negative result for coombs test until six months after passive immunization with investigational product.

SECONDARY OUTCOMES:
Adverse Events Report | up to six months
  Safety of human immunoglobulin anti-RhD will be verified through adverse events reported by participants throughout study. The adverse events will be classified about the type, frequency, intensity, seriousness, severity and relation to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Regina M Doi, physician, Study Director — Azidus Brasil Scientific Research and Development Ltda
Locations (5):
- Brazil (5):
  - Centro de Pesquisa da MEAC - Maternidade Escola Assis Chateaubriand, Fortaleza, Ceará
  - Instituto Tropical de Medicina Reprodutiva e Menopausa -INTRO, Cuiabá, Mato Grosso
  - Associação Educadora São Carlos AESC - Centro de Pesquisa HRPC, Canoas, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas (Puc-Rs), Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided